CLINICAL TRIAL: NCT05444218
Title: Clinical and Microbiological Effects of Surgical Access Combined With Systematically Administered Antibiotics in the Treatment of Peri-implantitis: 1-year Randomized Double-blinded Controlled Clinical Trial
Brief Title: Surgical Access Combined With Systematically Administered Antibiotics in the Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guarulhos (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Principal Investigator, Jamil awad shibli, Professor, University of Guarulhos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 40892620.9.0000.5506; 1454_2019 (Other: ITI Research Grant)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; open flap debridement; Er:YAG irradiation; metronidazole; amoxicillin; microbiota
MeSH Terms: conditions — Peri-Implantitis | interventions — Metronidazole; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Open flap debridement + Er: YAG irradiation alone + systemic placebo of metronidazole and amoxicillin thrice a day (TID) for 14 days
  Interventions: Procedure: Open flap debridement; Other: Er: YAG irradiation; Drug: Placebos
- Test (Experimental): Open flap debridement + Er: YAG irradiation alone + systemic metronidazole (400mg) and amoxicillin (500mg) thrice a day (TID) for 14 days
  Interventions: Procedure: Open flap debridement; Other: Er: YAG irradiation; Drug: Metronidazole; Drug: Amoxicillin

INTERVENTIONS:
Procedure: Open flap debridement — After local anesthesia (2% lidocaine with1:100,000 epinephrine), intrasulcular incisions will be performed to create a horizontal flap extending beyond the adjacent teeth and/or implants. Buccal and lingual full-thickness flaps will be dissected, and granulation tissue will be removed to expose the implant threads and bone defect. The flap will be repositioned in its original position and stabilized with interrupted sutures, which will be removed after 10 days.
  Other Names: OFD
Other: Er: YAG irradiation — An Er:YAG laser (Lite Touch, Light Instruments, Israel) will be used, with an irradiation energy of 20 mJ, frequency of 20 Hz, output power of 0.4 W, and an energy density of 2.76 J/cm2. An 8 mm long sapphire tip will be used in the respective handpiece and not in contact with the titanium surface, with concomitant water spray irrigation, under air 6 and water spray 6, the irradiation angle will be 90 degrees, at a focal distance of 2 mm, with spot size diameter of 1.3 mm
Drug: Metronidazole — Metronidazole 400 mg thrice a day for 14 days in the active phase of the periodontal treatment (beginning after open flap debridement).
  Other Names: MTZ
  Arms: Test
Drug: Amoxicillin — Amoxicillin 500 mg thrice a day for 14 days in the active phase of the periodontal treatment (beginning after open flap debridement).
  Other Names: AMX
  Arms: Test
Drug: Placebos — Amoxicillin and metronidazole placebos thrice a day for 14 days in the healing phase (beginning after open flap debridement).
  Arms: Control

SUMMARY:
This randomized clinical trial evaluates the clinical and microbiological (microbial complexes and changes in the diversity of the submucosal biofilm) effects of MTZ+AMX as adjuncts to anti-infectious surgical treatment plus Er: YAG in the treatment of peri-implantitis.

DETAILED DESCRIPTION:
Peri-implantitis is a pathological condition characterized by inflammation of peri-implant connective tissues and progressive peri-implant bone. Recently, the therapeutic protocol using non-surgical debridement associated with the combination of systemic metronidazole (MTZ) and amoxicillin (AMX) has not been shown to be effective in controlling the disease. These unfavorable results may have occurred due to the limitation in the change of the submucosal microbiological profile due to mechanical difficulties in the decontamination of the implant threads. Therefore, this randomized clinical trial (RCT) aimed to evaluate the clinical and microbiological (microbial complexes and changes in the diversity of the submucosal biofilm) effects of MTZ+AMX as adjuncts to anti-infectious surgical treatment plus Er:YAG in the treatment of peri-implantitis. Ninety-four subjects with untreated peri-implantitis are being included and will be randomly assigned to receive (i) open flap debridement plus Er:YAG irradiation alone (control), or (ii) with adjunctive systemically administered MTZ (400 mg) + AMX (500 mg) thrice a day (TID) for 14 days (test). Subjects will be monitored up to 12 months post-treatment. Submucosal biofilm samples from the deepest site of each implant with peri-implantitis will be collected in duplicate per patient: at baseline and at 3, 6 and 12 months post-therapy and analyzed by checkerboard DNA-DNA hybridization for 40 bacterial species, and at baseline, 3 and 12 months post-treatment for 16S rRNA sequencing (Ion Torrent PGM System). The primary outcome variable of this trial will be the difference between treatment groups for the change in CAL from baseline to 12 months. The significance of differences in each group (over the course of the study) will be sought using the Student's-t test; and among groups (at each time point) using either ANOVA /ANCOVA or Kruskal Wallis tests and post-hoc analyses, depending on normality of the data. Fisher's exact test will be used to compare differences in the frequency of gender. Statistical significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age;
* in general good health,
* at least one dental implant in function for at least one year with untreated peri-implantitis defined as: presence of bleeding and/or suppuration on gentle probing, probing depths (PD) ≥ 6mm, and bone levels ≥3mm apical of the most coronal portion of the intraosseous part of the implant.

Exclusion Criteria:

* subjects with ≥6 sites with PD ≥5mm;
* individuals that received periodontal treatment within three months prior to entering the study;
* inability to perform proper supramucosal and supragingival plaque control (e.g., due to improper restoration design or lack of skills);
* poorly adapted implant-supported restoration;
* diabetes;
* pregnancy;
* nursing;
* history of allergies to metronidazole and/or amoxicillin, or any other ingredient of oral care products;
* alcohol or drug abuse;
* any systemic diseases that could affect post-operative healing or that required antibiotic premedication for routine dental therapy;
* long-term use of mouthrinses;
* anti-inflammatory medications;
* any other drug that could interfere with the study outcomes within three months prior to entering the study;
* use of antibiotics within six months prior to entering the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Difference between treatment groups for the change in the clinical attachment level (CAL). | 12 months.

SECONDARY OUTCOMES:
Percentage of patients (and implants) reaching the following clinical endpoint for treatment: PD< 5mm, absence of BOP and no further bone loss. | 12 months.
Mean plaque index. | Baseline, 3, 6 and 12 months.
Mean gingival index. | Baseline, 3, 6 and 12 months.
Percentage of sites with bleeding on probing. | Baseline, 3, 6 and 12 months.
Percentage of sites with suppuration. | Baseline, 3, 6 and 12 months.
Probing depth. | Baseline, 3, 6 and 12 months.
Occurrence of headache obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of vomiting obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of diarrhea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of metallic taste obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of nausea obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Occurrence of irritability obtained through a questionnaire of adverse effects. | 14 days after taking antibiotic.
Proportions of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months.
Counts of periodontal pathogenic bacterial species. | Baseline, 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Shibli, Professor, Principal Investigator — University of Guarulhos
Locations (1):
- University of Guarulhos, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S313-S318. doi: 10.1002/JPER.17-0739. PMID 29926955
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Dreyer H, Grischke J, Tiede C, Eberhard J, Schweitzer A, Toikkanen SE, Glockner S, Krause G, Stiesch M. Epidemiology and risk factors of peri-implantitis: A systematic review. J Periodontal Res. 2018 Oct;53(5):657-681. doi: 10.1111/jre.12562. Epub 2018 Jun 7. PMID 29882313
- [Background] Shibli JA, Melo L, Ferrari DS, Figueiredo LC, Faveri M, Feres M. Composition of supra- and subgingival biofilm of subjects with healthy and diseased implants. Clin Oral Implants Res. 2008 Oct;19(10):975-82. doi: 10.1111/j.1600-0501.2008.01566.x. PMID 18828812
- [Background] Perez-Chaparro PJ, Duarte PM, Shibli JA, Montenegro S, Lacerda Heluy S, Figueiredo LC, Faveri M, Feres M. The Current Weight of Evidence of the Microbiologic Profile Associated With Peri-Implantitis: A Systematic Review. J Periodontol. 2016 Nov;87(11):1295-1304. doi: 10.1902/jop.2016.160184. Epub 2016 Jul 15. PMID 27420109
- [Result] Faggion CM Jr, Listl S, Fruhauf N, Chang HJ, Tu YK. A systematic review and Bayesian network meta-analysis of randomized clinical trials on non-surgical treatments for peri-implantitis. J Clin Periodontol. 2014 Oct;41(10):1015-25. doi: 10.1111/jcpe.12292. Epub 2014 Aug 11. PMID 25039292
- [Result] Swider K, Dominiak M, Grzech-Lesniak K, Matys J. Effect of Different Laser Wavelengths on Periodontopathogens in Peri-Implantitis: A Review of In Vivo Studies. Microorganisms. 2019 Jun 29;7(7):189. doi: 10.3390/microorganisms7070189. PMID 31261945
- [Result] Aoki A, Mizutani K, Schwarz F, Sculean A, Yukna RA, Takasaki AA, Romanos GE, Taniguchi Y, Sasaki KM, Zeredo JL, Koshy G, Coluzzi DJ, White JM, Abiko Y, Ishikawa I, Izumi Y. Periodontal and peri-implant wound healing following laser therapy. Periodontol 2000. 2015 Jun;68(1):217-69. doi: 10.1111/prd.12080. PMID 25867988
- [Result] Shibli JA. Is Laser the Best Choice for the Treatment of Peri-Implantitis? Photomed Laser Surg. 2018 Nov;36(11):569-570. doi: 10.1089/pho.2018.4521. No abstract available. PMID 30422756
- [Result] Feres M, Figueiredo LC, Soares GM, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015 Feb;67(1):131-86. doi: 10.1111/prd.12075. PMID 25494600
- [Result] Feres M, Retamal-Valdes B, Fermiano D, Faveri M, Figueiredo LC, Mayer MPA, Lee JJ, Bittinger K, Teles F. Microbiome changes in young periodontitis patients treated with adjunctive metronidazole and amoxicillin. J Periodontol. 2021 Apr;92(4):467-478. doi: 10.1002/JPER.20-0128. Epub 2020 Oct 12. PMID 32844406
- [Result] Teughels W, Feres M, Oud V, Martin C, Matesanz P, Herrera D. Adjunctive effect of systemic antimicrobials in periodontitis therapy: A systematic review and meta-analysis. J Clin Periodontol. 2020 Jul;47 Suppl 22:257-281. doi: 10.1111/jcpe.13264. PMID 31994207
- [Result] Shibli JA, Ferrari DS, Siroma RS, Figueiredo LC, Faveri M, Feres M. Microbiological and clinical effects of adjunctive systemic metronidazole and amoxicillin in the non-surgical treatment of peri-implantitis: 1 year follow-up. Braz Oral Res. 2019 Sep 30;33(suppl 1):e080. doi: 10.1590/1807-3107bor-2019.vol33.0080. eCollection 2019. PMID 31576959
- [Result] Tamashiro NS, Duarte PM, Miranda TS, Maciel SS, Figueiredo LC, Faveri M, Feres M. Amoxicillin Plus Metronidazole Therapy for Patients with Periodontitis and Type 2 Diabetes: A 2-year Randomized Controlled Trial. J Dent Res. 2016 Jul;95(7):829-36. doi: 10.1177/0022034516639274. Epub 2016 Mar 24. PMID 27013640
- [Result] Borges I, Faveri M, Figueiredo LC, Duarte PM, Retamal-Valdes B, Montenegro SCL, Feres M. Different antibiotic protocols in the treatment of severe chronic periodontitis: A 1-year randomized trial. J Clin Periodontol. 2017 Aug;44(8):822-832. doi: 10.1111/jcpe.12721. Epub 2017 Jul 26. PMID 28303587
- [Result] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807